CLINICAL TRIAL: NCT02235519
Title: A Randomized, Open Label Study to Evaluate the Pleiotropic Effects of Azilsartan Medoxomil 40 and 80 mg for 12 Weeks Over Metabolic Markers in Patients With Hypertension, Obesity or Type 2 Diabetes Mellitus
Brief Title: Pleiotropic Effects of Azilsartan Medoxomil Over Insulin Resistance in Obese, Diabetic and Hypertensive Patients
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital General de México Dr. Eduardo Liceaga (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DI/12/404B/4/85
Record Dates: First submitted 2014-09-05; First posted 2014-09-10 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2014-09

CONDITIONS: Hypertension; Obesity; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Hypertension; Obesity; Diabetes Mellitus, Type 2 | interventions — azilsartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Azilsartan low dosage (Active Comparator): Patients will take azilsartan 40 mg during 12 weeks
  Interventions: Drug: Azilsartan 40 mg.
- Azilsartan high dosage (Active Comparator): Patients will take azilsartan 80 mg during 12 weeks
  Interventions: Drug: Azilsartan 80 mg

INTERVENTIONS:
Drug: Azilsartan 40 mg. — Patients will take 40 mg of azilsartan during 12 weeks
  Other Names: Edarbi 40 mg
  Arms: Azilsartan low dosage
Drug: Azilsartan 80 mg — Patients will take 80 mg of azilsartan during 12 weeks
  Other Names: Edarbi 80 mg
  Arms: Azilsartan high dosage

SUMMARY:
The goal of this study is to build a mathematical model to explain the effect of two doses of azilsartan (40 and 80 mg) upon metabolic (insulin resistance, glucose) and inflammatory parameters (cytokines) in function of "metabolic strata" like obesity, type 2 diabetes mellitus, hypertension and their combinations.

DETAILED DESCRIPTION:
There are data supporting angiotensin II receptor subtype 1 (AT1) antagonist have beneficial effects on metabolic control due to some pleiotropic effect mediated by peroxisome proliferator-activated receptor (PPAR) gamma induction. Azilsartan is a prodrug absorbed in the gastrointestinal tract that can improve metabolic milieu under diverse conditions like obesity, hypertension (can be considered a metabolic disease) or type 2 diabetes mellitus. Clinical studies that have been raised in this regard are few, and still show controversial issues.

The objective of any study with AT1 antagonist drug interested in pleiotropic effects should not only focus on antihypertensive improvement, but also the effect on other areas such as metabolism of lipids and carbohydrates in obese and/or type 2 diabetes.

This study is a randomized, open labeled, clinical study. The aim is to build a mathematical model for supporting the effect of azilsartan 40 or 80 mg on metabolic and inflammatory measurements in function of metabolic conditions (i.e. obesity, type 2 diabetes and hypertension, and their combinations).

Patients will be stratified according to their metabolic status and randomized by blocks of four for each strata. This strategy will help to maintain each treatment group in balance. All subjects will receive the treatment for 12 weeks.

Subjects who attend the outpatient consultation at the Hospital General de Mexico will be invited to participate in the study. Those who meet the inclusion criteria must sign an informed consent approved by the ethics committee. This document describes the follow-up visits as described below:

Screening visit (V-1):

This visit includes patient history, physical examination (weight, height, waist circumference and blood pressure) and a blood sample for measurement of: complete blood count, fasting glucose, HbA1c, creatinine, adiponectin, IL-1b, IL-6, IL-10, TNF-α, liver function tests, C-reactive protein, blood chemistry, proteinuria, 24-hours urinary glucose and creatinine.

Initial visit (V0):

Physical examination will be performed and blood samples for oral glucose tolerance test will be drawn at 0, 30, 60, 90 and 120 minutes, with these data points the Matsuda insulin sensitivity index will be calculated. Pharmacological treatment of 40mg or 80mg azilsartan 4 weeks will be assigned (open labeled but randomized).

Visit 1 and 2 (V1, V2):

These visits performed at 4 and 8 weeks respectively include: physical examination, recording of adverse events and medication count to check adherence to treatment accomplishment.

Visit 3 (V3):

Week 12 include physical examination, adverse events registration, complete blood count, fasting glucose, HbA1c, creatinine, adiponectin, IL-1b, IL-6, IL-10, TNF - α, liver function tests, C reactive protein, blood chemistry, proteinuria, 24-hours urinary glucose and creatinine. Furthermore an oral glucose tolerance test with samples at 0, 30, 60, 90 and 120 minutes will be taken, to calculate the index of insulin sensitivity by the Matsuda method.

Statistical analysis and sample size. The sample size was calculated for ANCOVA analysis considering 8 groups with 5 covariates. Considering an alpha error of 5%, effect size of 30%, and statistical power of 90% a total sample of 250 patient was calculated. If we consider a 20% attrition of the sample, giving a total of 300 patients, i.e. 150 patients per treatment group.

A descriptive analysis will be done. The contrast among groups will be analyzed by an ANCOVA model and the function fitness will be calculated using ordinary least squares. Dependent variables will be insulin sensitivity, proteinuria, stiffness of the carotid artery, cytokines. Fixed factors: sex, blood pressure category, metabolic status, drug treatment. Covariates: Age, waist circumference.

The greatest expected size of effect would be within the group of patients with obesity, hypertension, and type 2 diabetes mellitus (all three) treated with 80 mg and the lowest size of effect within the group of only obesity treated with 40 mg.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent in accordance with Good Clinical Practices and local legislations
2. Age between ≥25 and ≤ 65 years
3. Patients with hypertension stage 1 as defined by systolic blood pressure (SBP) ≥140 but <159 mmHg and diastolic blood pressure (DBP) ≥90 but < 99 mmHg at randomization
4. Ability to stop any current antihypertensive therapy without unacceptable risk to the patient (Investigator's discretion)
5. BMI ≥25 and ≤35.
6. Patients with type 2 diabetes mellitus can participate and will be stratified before randomization. Diagnosis can be established by clinical history, 75-g oral glucose tolerance test (ADA criteria), or fasting glucose > 126 mg/dL.

Exclusion Criteria:

1. Pre-menopausal women (last menstruation ≤1 year prior to signing informed consent) who are not surgically sterile, nursing, are pregnant or without any anticonceptive methods.
2. Known hypersensitivity to the study drug
3. Gastrointestinal surgery which might alter absorption, distribution, or drug metabolism.
4. History of angioedema related to ACE inhibitors or angiotensin II receptor blockers.
5. Night shift workers who routinely sleep during the daytime and whose work hours include midnight to 4:00 a.m.
6. Known or suspected secondary hypertension (e.g., renal artery stenosis or phaeochromocytoma)
7. SBP≥160 mmHg and/or DBP ≥100 mmHg
8. Renal dysfunction as defined by: serum creatinine >3.0 mg/dL (or >265 umol/L) and/or creatinine clearance <30 ml/min and/or other clinical markers of severe renal impairment.
9. Bilateral renal arterial stenosis, renal artery stenosis in a solitary functional kidney, post-renal transplant patients or patients with one kidney
10. Clinically relevant hypokalemia or hyperkalemia (i.e., <3.5 mmol/L or >5.5 mmol/L, may be rechecked for suspected error in result)
11. Uncorrected sodium or volume depletion
12. Primary aldosteronism.
13. Hereditary fructose intolerance
14. Biliary obstructive disorders (e.g., cholestasis) or hepatic insufficiency
15. Congestive heart failure class III-IV according to criteria fron the New York Heart Association.
16. Clinically significant ventricular tachycardia, atrial fibrillation, atrial flutter or other clinically relevant cardiac arrhythmias as determined by the Investigator.
17. Hypertrophic obstructive cardiomyopathy, severe obstructive coronary artery disease, aortic stenosis, hemodynamically relevant stenosis of the aortic or mitral valve
18. Patients whose diabetes has not been stable and controlled for at least the past 3 months as defined by an Glycosylated Hemoglobin A1c >=10% or fasting glucose greater than 400 mg/dL.
19. Patients who have previously experienced symptoms characteristic of angioedema during treatment with ACE inhibitors or angiotensin-II receptor antagonists
20. History of drug or alcohol dependency within 6 months prior to signing the informed consent form
21. Concomitant administration of any medications known to affect blood pressure, except medications allowed by the protocol
22. Any investigational drug therapy within 1 month of signing the informed consent
23. Known hypersensitivity to any component of the trial drugs (telmisartan, hydrochlorothiazide, or placebo)
24. History of non-compliance or inability to comply with prescribed medications or protocol procedures (less than 80% or more than 120%, especially during run-in).
25. Any other clinical condition which, in the opinion of the investigator, would not allow safe completion of the protocol and safe administration of the trial medication

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Blood pressure | 12 weeks
  Effect size of azilsartan medoxomil 40 and 80 mg in lowering systolic and diastolic blood pressure stratified by metabolic condition (obesity or type 2 diabetes mellitus). The minimal size effect between groups will be at least 30% and absolute percentage of previous hypertensive subjects reaching targeted values of < 130/85 mmHg.

SECONDARY OUTCOMES:
Insulin sensitivity and HbA1c level | 12 weeks
  Effect over insulin sensitivity measured by Matsuda index of insulin sensitivity (ISI) and the level of HbA1c. The function will show a increase for ISI that in a within contrast will be larger for those with obesity with hypertension and diabetes. Meanwhile the HbA1 will show a deep decrease for the same group.
Effect of azilsartan on Inflammatory markers | 12 weeks
  Effect size between azilsartan 40 mg and 80 mg on inflammatory markers (IL-1b, IL-6, IL 10, TNF-α, and adiponectin). A decrease in this response will be more important for the 80 mg and those with obesity, hipertension and diabetes.
Endothelial function | 12 weeks
  Subjects with stiffness of the carotid and brachial artery will show improvement in relaxation, and the larger effect will be for 80 mg in the group of obesity, hypertension and diabetes mellitus.
Renal function improvement. | 12 weeks
  Proteinuria will show a significant decrease after 12 weeks of treatment with azilsartan. The larger effect will be for the 80 mg and the obese, hypertension and diabetic group.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Peralta, MD, Principal Investigator — HGM; Rogelio Zapata, MD, Study Chair — HGM; Estrella Martinez, RN, Study Director — HGM
Locations (1):
- Hospital General de Mexico "Dr. Eduardo Liceaga", Mexico City, Mexico City, Mexico